CLINICAL TRIAL: NCT05816122
Title: MS-DETECT: Early Detection of Multiple Sclerosis Progression With MSCopilot® Detect
Acronym: MS-DETECT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ad scientiam (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MS-DETECT
Record Dates: First submitted 2023-03-13; First posted 2023-04-18 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- MSCopilot® Detect (Experimental): Performance of digital tests and standard test in clinic at D0, M6, M12, M18 and M24 (if applicable) Use of MSCopilot® Detect at-home in between visits during 18 or 24 months (if applicable)
  Interventions: Device: MSCopilot® Detect mobile application

INTERVENTIONS:
Device: MSCopilot® Detect mobile application — MSCopilot® Detect includes active tests for walking, cognition, dexterity and vision, and e-questionnaires related to fatigue and Multiple Sclerosis quality of life

SUMMARY:
The study aims to evaluate MSCopilot® Detect, a smartphone application for at-home monitoring of patients with Multiple Sclerosis (MS).

The primary objective is to enhance and standardize remote monitoring of MS patients to accurately assess disease progression caused by either Relapse Activity Worsening (RAW) or Progression Independent of Relapses (PIRA). The study also aims to assess the safety, usability, and satisfaction of the solution.

A secondary objective is to determine MSCopilot® Detect's ability to provide early detection of disease changes and predict changes in Expanded Disability Status Scale (EDSS) scores in more patients.

Exploratory objectives include evaluating the relationship between MSCopilot® Detect composite and individual scores and other biomarkers such as MRI, soluble glial fibrillary acidic protein (sGFAP), and soluble neurofilament light chain (sNfL).

Patients will be able to download the free MSCopilot® Detect app. They will participate in 1 inclusion visit and 3 follow-up visits, scheduled at 6 months, 12 months, and 18 months (an additional visit at 24 months may be scheduled if necessary). Every 3 months, patients will complete validated questionnaires regarding MS symptoms and quality of life and participate in digital tests designed to monitor MS symptom progression.

The study will include 336 MS patients and will be conducted in the United States, Canada, Germany, Italy, Spain, Denmark and France

ELIGIBILITY:
Inclusion Criteria:

* Adult patients living with RRMS or SPMS, aged 30 to 65
* EDSS score between 2.5 to 6.5 points
* With a disease duration > 5 years
* Clinically stable during the last 3 months before inclusion (no relapses, no disability progression)
* No change in the DMT* during the last 3 months before inclusion
* Receiving optimal symptomatic treatments at baseline (clinician's judgment)
* Owns a personal smartphone which mobile operating system is above 14 for IOS (iPhone) and 8 for Android included with a good internet connexion
* Able to use a smartphone
* Able to read language in wich the mobile application is available and able to understand pictograms.
* Applicable to patients enrolled in France only: affiliated to a social security system.

Exclusion Criteria:

* Medically unstable conditions that may hinder patient's ability to comply with the study procedures
* Inability to use a smartphone or MSCopilot® Detect application
* Patient with corrected visual acuity less than 4/10 (Monoyer) or 20/50 (Snellen at 20 feet) or +0,4 (LogMAR)
* Pregnancy and nursing women
* Persons under guardianship or curatorship
* Current drugs or/and alcohol abuse that could influence performance on the tests (clinician's judgment)
* Patients have participated in another clinical study within the previous 30 days of screening or are currently participating in another study that, in the opinion of the Investigator, might interfere with the patient's full participation in the study or confound the assessment of the patient or outcome of the study.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate MSCopilot® Detect individual scores and/or composite scores sensitivity to detect disability worsening based on revised-MSFC scores. | Throughout the study at each hospital visit: Day 0, Month 6, Month 12, Month 18 and Month 24 (if applicable)
  The discriminatory ability of the MSCopilot® Detect application in detecting clinically meaningful worsening (disability worsening) based on the revised-MSFC will be evaluated using the Area Under the ROC Curve (AUC) method. Confidence intervals will also be estimated.
  The minimum significant AUC value will be set at >0.67, and Confidence Intervals will be calculated. Sensitivity and specificity will also be determined. To validate the estimated AUC values and cutoffs generated by the MSCopilot® Detect application, a train/test set will be utilised.

SECONDARY OUTCOMES:
To evaluate MSCopilot® Detect individual scores and/or composite scores sensitivity to detect disability worsening based on EDSS. | Throughout the study at each hospital visit: Day 0, Month 6, Month 12, Month 18 and Month 24 (if applicable)
  The study will evaluate the sensitivity, specificity, concordance, and accuracy of the MSCopilot® Detect application in predicting confirmed disability worsening (CDW) at 24 weeks as also captured by the EDSS, using a contingency table.
  We will also generate time series box plots of MSCopilot® Detect individual scores and/or composite scores based on the patient progression status (determined by EDSS), using both intra-patient and inter-patient visualisation.
To evaluate MSCopilot® Detect individual scores and/or composite scores sensitivity to detect disability worsening earlier than the EDSS. | Throughout the study at each hospital visit: Day 0, Month 6, Month 12, Month 18 and Month 24 (if applicable)
  The time to progression-free events based on EDSS and MSCopilot® Detect individual scores and/or composite scores will be estimated with a Kaplan-Meier method (Log-rank test for comparison). Univariate and multivariate survival models (e.g. Cox or Anderson-Gill survival model), will be used to estimate Hazards Rates (HRs), if relevant.
  Proportions of disability worsening based on MSCopilot® Detect composite or individual scores and worsening based on the EDSS 24-week CDW will be compared for each timepoint.
  Time series boxplot of MSCopilot® Detect individual scores and/or composite score according to the patient disability worsening (by EDSS) intra-patient and inter-patient.
To evaluate MSCopilot® Detect individual and/or composite scores ability to detect disease progression in absence of a relapsing activity (PIRA). | Throughout the study at each hospital visit: Day 0, Month 6, Month 12, Month 18 and Month 24 (if applicable)
  Proportion of patients with PIRA (progression independent of relapses) based either on EDSS 24-week CDP compared to the proportion of patients with PIRA based on MSCopilot® Detect composite or individual scores progression status.
To evaluate MSCopilot® Detect individual scores and/or composite scores ability to detect MSFC changes over time. | Throughout the study at each hospital visit: Day 0, Month 6, Month 12, Month 18 and Month 24 (if applicable)
  Slopes parameters will be computed using a mix model to characterize the change from baseline in MSCopilot® Detect individual and/or composite scores and revised-MSFC scores over time.
  The association between these slopes parameters will be assessed using correlation coefficient.
To measure MSCopilot® Detect individual scores and/or composite scores association with the clinical scores. | Throughout the study at each hospital visit: Day 0, Month 6, Month 12, Month 18 and Month 24 (if applicable)
  The association between digital and clinical scores will be studied with correlation coefficient calculated between:
  * MSCopilot® Detect individual scores ((MWPT, MDT, MCT, MVT and Mobile Walking Endurance Test (MWET)) and/or composite score at home and EDSS score performed in clinic.
  * MSCopilot® Detect individual scores (MWPT, MDT, MCT, MVT and MWET) and/or composite score at home and revised-MSFC-3 or Revised-MSFC3 + SLCLAT scores performed in clinic.
To assess reproducibility of MSCopilot® Detect individual scores and/or composite scores between in-clinic and at-home digital tests. | At home (Day 1, Month 6+1 day, Month 12 + 1 day, Month 18-1 day and Month 24-1 day (if applicable)) and in-clinic ((Day 0, Month 6, Month 12, Month 18 and Month 24 (if applicable))
  Intraclass correlation coefficient (ICC) between MSCopilot® Detect individual scores and/or composite score at home and in-clinic.
To assess reliability of MSCopilot® Detect individual scores and/or composite scores at-home over time. | Day 0 versus Month 6, Month 6 versus Month 12, Month 12 versus Month 18, Month18 versus Month 24 (if applicable) AND Day 0 to Month 18 or Day 0 to Month 24 (if applicable) and Day 0 to Month 15 or Day 0 to Month 21 (if applicable) at home.
  Intraclass correlation coefficient (ICC) of MSCopilot® Detect individual scores and/or composite score at home with a maximum paired time point of 6 months.
  ICC of MSCopilot® Detect individual scores and/or composite score at home will over time.
To evaluate Patient QoL (Multiple Sclerosis Impact Scale: MSIS-29 and Modified Fatigue Impact Scale - 5-item version: MFIS-5) and their association with MSCopilot® Detect individual and composite scores. | Throughout the study between in clinic visit, an average of 24 months
  Analysis of MSIS-29 and MFIS-5 questionnaires:
  Descriptive analysis of questionnaire scores over time. Comparison of Patient QoL between patients with and without a confirmed disability worsening Correlation between MSCopilot® Detect individual and/or composite score at home and Questionnaires scores (MSIS29 and MFIS-5).
  Sensitivity, specificity, concordance, and accuracy will be evaluated between clinically meaningful change of MSCopilot® Detect application (individual and composite scores) and questionnaires (MSIS29 and MFIS-5).
  Proportions comparison of patients with a clinically meaningful change will be assessed between MSCopilot® Detect application (individual and composite scores) and questionnaires (MSIS29 and MFIS-5).
  Clinically meaningful change for questionnaires:
  MSIS-29: 8-point change compared to baseline. MFIS-5: 4-point change compared to baseline.
To evaluate the ability of MSCopilot® Detect individual scores and/or composite score to discriminate between a relapse and a momentary disability worsening (+1 point EDSS score for an initial EDSS <5,5; +0.5 point for an initial EDSS ≥5.5). | Throughout the study at each hospital visit: Day 0, Month 6, Month 12, Month 18 and Month 24 (if applicable)
  Descriptive analysis:
  MSCopilot® Detect individual and/or composite score profiles, between relapse and a momentary disability worsening patient.
  Annualized Relapse Rate (ARR) calculation. Logistic regression to estimate Area under ROC Curve (i.e. discriminatory power).
To evaluate MSCopilot® Detect Safety | Throughout the study between in clinic visit, an average of 24 months
  Descriptive analysis of the number of Adverse Events related to MSCopilot® Detect will be reported.
To evaluate MSCopilot® Detect Adherence | Throughout the study between in clinic visit, an average of 24 months
  Descriptive analysis of the mobile application's adherence data (number of completed questionnaires, number of performed tests, number of performed sessions, etc.)
To assess the satisfaction and user experience with the MSCopilot® Detect smartphone application and the MSCopilot® Detect web dashboard. | Every 3 months for about 24 months
  Descriptive analysis over the course of the study of the answers to the patient satisfaction and user experience questionnaires related to the use of the MSCopilot® Detect smartphone application.
To assess the satisfaction and user experience with the MSCopilot® Detect web dashboard. | Every 6 months for about 24 months
  Descriptive analysis over the course of the study of the answers to physician satisfaction & user experience questionnaires relative to the use of the MSCopilot® Detect web dashboard.
To describe the evolution of MSCopilot® Detect individual scores and/or composite scores at-home over time. | Throughout the study between in clinic visit, an average of 24 months
  The time to progression-free events based on MSCopilot® Detect individual scores and/or composite scores will be estimated with a Kaplan-Meier method (Log-rank test for comparison). Univariate and multivariate survival models (e.g. Cox or Anderson-Gill survival model), will be used to estimate Hazards Rates (HRs), if relevant.
  Cumulative proportions of disability worsening based on MSCopilot® Detect composite or individual scores for each timepoint.
  Time series boxplot of MSCopilot® Detect individual scores and/or composite score according to the patient disability worsening (by MSCopilot® Detect) using both intra-patient and inter-patient visualisation.

CONTACTS AND LOCATIONS:
Locations (34):
- United States (10):
  - Jennifer Graves, San Diego, California
  - Joash Lazarus Sr., Atlanta, Georgia
  - Daniel Wynn, Northbrook, Illinois
  - Craig E. Herrman, Indianapolis, Indiana
  - Jennifer Feng, New Orleans, Louisiana
  - Robert Naismith, St Louis, Missouri
  - Aaron Boster, Columbus, Ohio
  - Gabriel Pardo, Oklahoma City, Oklahoma
  - Vijayshree Yadav, Portland, Oregon
  - Leorah Freeman, Austin, Texas
- Canada (4):
  - Galina Vorobeychik, Burnaby
  - Mark Freedman, Ottawa
  - St. Michael's Hospital, Toronto
  - Robert Carruthers, Vancouver
- Denmark (3):
  - University Hospital of Southern Denmark, Esbjerg
  - Finn Sellebjerg, Glostrup Municipality
  - Sivagini Prakash, Viborg
- France (5):
  - Hôpital Roger Salengro, Lille
  - Cécile Donzé, Lomme
  - Adil Maarouf, Marseille
  - Mikael Cohen, Nice
  - Bertrand Bourre, Rouen
- Germany (3):
  - Boris-Alexander Kallman, Bayreuth
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Rupert Knoblich, Erbach im Odenwald
- Italy (3):
  - Emilio Portaccio, Florence
  - Emanuele D'Amico, Foggia
  - IRCCS Ospedale San Raffaele, Milan
- Spain (6):
  - Gary Álvarez Bravo, Girona
  - Enric Monreal, Madrid
  - University Hospital San Carlos, Madrid
  - Ana Alonso, Málaga
  - Miguel Llaneza, Oviedo
  - Jesùs Martin, Zaragoza

IPD SHARING:
Plan to Share IPD: No